CLINICAL TRIAL: NCT02432404
Title: Effects of a Vaginal Contraceptive Ring on Vaginal Microbiota and Local Immunity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Christine Johnston, Assistant Professor, Medicine/Division of Allergy and Infectious Diseases, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003584; U19AI113173 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-05-04 (Estimated); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Bacterial Vaginosis
Keywords: HSV-2; Contraceptive Vaginal Ring
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclic NuvaRing CVR Use (Active Comparator): CVR use for 3 weeks, remove for 1 week, then replace
  Interventions: Drug: NuvaRing
- Continuous NuvaRing CVR Use (Experimental): CVR use for 4 weeks, then replace
  Interventions: Drug: NuvaRing

INTERVENTIONS:
Drug: NuvaRing

SUMMARY:
To assess potential benefits associated with both intermittent (use for 3 weeks, remove for 1 week, as defined in the package insert) and continuous (use for 4 weeks, then replace) CVR use among women either with BV or at high risk for BV. The investigators will also recruit women who are HSV2-infected.

ELIGIBILITY:
Inclusion Criteria:

* ≥18-40 year old women
* BV+ by Amsel criteria and Nugent score OR history of BV in the prior 6 months
* Willing to use the NuvaRing as directed
* Not intending or wishing to become pregnant over the course of the study
* Capable of providing written informed consent

Exclusion Criteria:

* Current pregnancy
* Desire/intent to become pregnant over the course of the study
* Women who are less than 6 weeks postpartum
* Contraindications to hormonal contraceptive use per package insert, including history of deep vein thrombosis, smoking in women older than 35 years
* Current IUD
* Unable to comprehend consent material because of language barrier or psychological difficulty

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Johnston, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- UW Virology Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Background] Veres S, Miller L, Burington B. A comparison between the vaginal ring and oral contraceptives. Obstet Gynecol. 2004 Sep;104(3):555-63. doi: 10.1097/01.AOG.0000136082.59644.13. PMID 15339769
- [Background] Atashili J, Poole C, Ndumbe PM, Adimora AA, Smith JS. Bacterial vaginosis and HIV acquisition: a meta-analysis of published studies. AIDS. 2008 Jul 31;22(12):1493-501. doi: 10.1097/QAD.0b013e3283021a37. PMID 18614873
- [Background] Cohen CR, Lingappa JR, Baeten JM, Ngayo MO, Spiegel CA, Hong T, Donnell D, Celum C, Kapiga S, Delany S, Bukusi EA. Bacterial vaginosis associated with increased risk of female-to-male HIV-1 transmission: a prospective cohort analysis among African couples. PLoS Med. 2012;9(6):e1001251. doi: 10.1371/journal.pmed.1001251. Epub 2012 Jun 26. PMID 22745608
- [Background] Heffron R, Donnell D, Rees H, Celum C, Mugo N, Were E, de Bruyn G, Nakku-Joloba E, Ngure K, Kiarie J, Coombs RW, Baeten JM; Partners in Prevention HSV/HIV Transmission Study Team. Use of hormonal contraceptives and risk of HIV-1 transmission: a prospective cohort study. Lancet Infect Dis. 2012 Jan;12(1):19-26. doi: 10.1016/S1473-3099(11)70247-X. Epub 2011 Oct 3. PMID 21975269
- [Background] Vodstrcil LA, Hocking JS, Law M, Walker S, Tabrizi SN, Fairley CK, Bradshaw CS. Hormonal contraception is associated with a reduced risk of bacterial vaginosis: a systematic review and meta-analysis. PLoS One. 2013 Sep 4;8(9):e73055. doi: 10.1371/journal.pone.0073055. eCollection 2013. PMID 24023807

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After 1 month baseline observation, participants initiated the CVR and were followed monthly for 4 months
Groups:
- NuvaRing CVR Use: Participants could choose to use CVR for 3 weeks, remove for 1 week, then replace, or to use continuously.
  NuvaRing
Period: Overall Study
Arm/Group | NuvaRing CVR Use
Started | 81
Initiated Nuvaring CVR | 61
Completed | 45
Not Completed | 36

BASELINE CHARACTERISTICS:
Arm/Group | NuvaRing CVR Use
Number analyzed (Participants) | 81
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: 9 persons had missing age
  years
    number analyzed (Participants) | 72
    (all) | 28 [23 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported.
  In this analysis, participants selected "other" as a category. This will be indicated in the more than one race" count, since "other" is not available.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 23
    White | 38
    More than one race | 15
    Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 81

OUTCOME MEASURES:

1. Primary Outcome: Quantity of BV-associated Bacteria by qPCR and High-throughput Sequencing Tests
Description: Change in Log10 quantity of bacteria detected (L. crisptatus, L. jensenii, L. iners, G. vaginalis, Megasphaera spp. BVAB2)
Time Frame: Up to 8 months
Population: Participants who initiated the ring and had at least one followup month in M3/4/5/6
Measure: Mean (Standard Deviation); unit: log10 copies/ml
Units Other Than Participants: swabs
Groups:
- NuvaRing CVR Use: Participants could choose to use NuvaringCVR for 3 weeks, remove for 1 week, then replace, or to use continuously.
Arm/Group | NuvaRing CVR Use
Number analyzed (Participants) | 57
Number analyzed (swabs) | 2895
log10 copies/ml
  G. vaginalis Baseline (M1-M2) | 5.59 (2.27)
  G. vaginalis Nuvaring (M2-M3) | 5.22 (2.42)
  G. vaginalis Nuvaring (M3-M6) | 4.91 (2.13)
  L. iners Baseline (M1-M2) | 7.41 (2.80)
  L. iners Nuvaring (M2-M3) | 7.49 (2.90)
  L. iners Nuvaring (M3-M6) | 7.89 (2.32)
  L. crispatus Baseline (M1-M2) | 5.60 (3.42)
  L. crispatus Nuvaring (M2-M3) | 5.82 (3.42)
  L. crispatus Nuvaring (M3-M6) | 5.94 (3.05)
  L. jensenii Baseline (M1-M2) | 4.85 (2.74)
  L. jensenii Nuvaring (M2-M3) | 4.97 (2.76)
  L. jensenii Nuvaring (M3-M6) | 5.23 (2.27)
  Megasphaera Baseline (M1-M2) | 2.50 (1.70)
  Megasphaera Nuvaring (M2-M3) | 2.60 (1.83)
  Megasphaera Nuvaring (M3-M6) | 2.20 (0.87)
  BVAB2 Baseline (M1-M2) | 2.22 (1.27)
  BVAB2 Nuvaring (M2-M3) | 2.29 (1.17)
  BVAB2 Nuvaring (M3-M6) | 2.12 (0.56)
Statistical Analysis 1: Comparison: NuvaRing CVR Use; Mean quantity of G. vaginalis at baseline and during Nuvaring Use (M2-M3); Test type: Other; p = 0.011, Random effects mixed model — p<0.05 is considered statistically significant; Random effects mixed model: random effects for subject and time category, with unstructured covariance, and AR(1) residuals; and robust SEs; Mean Difference (Final Values) = -0.37
Statistical Analysis 2: Comparison: NuvaRing CVR Use; Mean quantity of G. vaginalis at baseline and during Nuvaring Use (M3-M6); Test type: Other; p = 0.008, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.69
Statistical Analysis 3: Comparison: NuvaRing CVR Use; Mean quantity of L. iners at baseline and during Nuvaring Use (M2-M3); Test type: Other; p = 0.662, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.08
Statistical Analysis 4: Comparison: NuvaRing CVR Use; Mean quantity of L. iners at baseline and during Nuvaring Use (M3-M6); Test type: Other; p = 0.41, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.48
Statistical Analysis 5: Comparison: NuvaRing CVR Use; Mean quantity of L. crispatus at baseline and during Nuvaring Use (M2-M3); Test type: Other; p = 0.164, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.23
Statistical Analysis 6: Comparison: NuvaRing CVR Use; Mean quantity of L. crispatus at baseline and during Nuvaring Use (M3-M6); Test type: Other; p = 0.183, Random effects mixed model — p<0.05 is considered statistically significant; Mean Difference (Final Values) = 0.35
Statistical Analysis 7: Comparison: NuvaRing CVR Use; Mean quantity of L. jensenii at baseline and during Nuvaring Use (M2-M3); Test type: Other; p = 0.506, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.12
Statistical Analysis 8: Comparison: NuvaRing CVR Use; Mean quantity of L. jensenii at baseline and during Nuvaring Use (M3-M6); Test type: Other; p = 0.119, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.38
Statistical Analysis 9: Comparison: NuvaRing CVR Use; Mean quantity of Megasphaera at baseline and during Nuvaring Use (M2-M3); Test type: Other; p = 0.510, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.10
Statistical Analysis 10: Comparison: NuvaRing CVR Use; Mean quantity of Megasphaera at baseline and during Nuvaring Use (M3-M6); Test type: Other; p = 0.168, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.30
Statistical Analysis 11: Comparison: NuvaRing CVR Use; Mean quantity of BVAB2 at baseline and during Nuvaring Use (M2-M3); Test type: Other; p = 0.454, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07
Statistical Analysis 12: Comparison: NuvaRing CVR Use; Mean quantity of BVAB2 at baseline and during Nuvaring Use (M3-M6); Test type: Other; p = 0.471, Random effects mixed model — p<0.05 is considered statistically significant; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.10

2. Secondary Outcome: Number of Visits With BV
Description: Number of visits with BV prior to use of NuvaRing CVR compared to during NuvaRing CVR use.
Time Frame: Up to 8 months
Population: Among participants who initiated the ring and had at least one followup month in M3/4/5/6
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | NuvaRing CVR Use
Number analyzed (Participants) | 57
Number analyzed (Visits) | 320
Visits
  Visits with BV pre-CVR | 15
  Visits with BV at M3 | 6
  Visits with BV at M4/5/6 | 4

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | NuvaRing CVR Use
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 8/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NuvaRing CVR Use (N=45)
Vulvovaginal candidiasis (Reproductive system and breast disorders) | 8 (8) — Number of participants with vulvovaginal candidiasis at Final study visit

LIMITATIONS AND CAVEATS:
High rate of participant withdrawal from the study Single center experience

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02432404/Prot_SAP_000.pdf